CLINICAL TRIAL: NCT04164589
Title: EFFECTIVENESS OF THE NEUROADAPTATIVE REGULATION TECHNIQUE FOR THE TREATMENT OF URGE INCONTINENCE AND MIXED INCONTINENCE
Brief Title: EFFECTIVENESS OF THE NEUROADAPTATIVE FOR URGE INCONTINENCE
Acronym: SCENAR-EC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Principe de Asturias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCENAR-EC
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: A randomized, single blind placebo controlled clinical trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The Neuro-Adaptative Regulation will be carried out in the regime of switched off power supply in vulvo-perineal and sacral area.
  Interventions: Device: SCENAR 1NT-02.2
- Experimental (Experimental): The neuro-adaptative regulation will be carried out in vulvo-perineal and sacarl area.
  Interventions: Device: SCENAR 1NT-02.2

INTERVENTIONS:
Device: SCENAR 1NT-02.2 — The neuro-adaptative regulation will be carried out in vulvo-perineal and sacral area
  Other Names: Neuro-adaptative regulation

SUMMARY:
In this clinical trials the sponsor want to assess a self-controlled-energo-neuroadaptative-regulation in patient with urge incontinence

DETAILED DESCRIPTION:
In this clinical trials the sponsor want to assess a self-controlled-energo-neuroadaptative-regulation in patient with urge incontinence and mixted incontinence

ELIGIBILITY:
Inclusion Criteria:

* Urge incontinence or mixed incontinence without urethral hypermobility
* Over 3 months of disease evolves.

Exclusion Criteria:

* Severe physical limitations that might interfere with applying the treatment.
* Severe mental disorders that need pharmacology treatments that may influence in neuronal activity
* Oncological processes in the lower abdomen that had required radical surgery.
* Neurogenic bladder.
* Blockage of the bladder
* Vaginal infection
* Bladder infection or disorder of kidney function
* Have received, in the last year, botulinum toxin in bladder or pelvic organs.
* Have received pharmacological treatment for urge incontinence in the last month (before entry date in the trial)
* Be receiving pharmacological treatment for urge incontinence.
* Stress incontinence due to urethral hypermobility which was treatable with surgery.
* Pregnant women
* Patients with pacemarker

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Resultant value achieved in the assessment scale of urge incontinence. | 2 years
  Resultant value achieved in the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF). The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence. Question items: Frequency or urinary incontinence; Amount of leakage; Overall impact of urinary incontinence; Self-diagnostic ítem. Scoring scale: 0-21. Higher score mean a worse outcome.
Sandvik Test for Urinary Incontinence | 2 years
  It is a severity indez score of symptoms to calculate severity of urinary incontinence in women. Scores are from 0 to 12. The higher score: the more severe the urinary incontinence.

SECONDARY OUTCOMES:
Intervals between voiding | 2 years
  time between voiding
Frequency of nocturia | 2 years
  Frequency of nocturia
Quality of life index (Potenziani-14-CI-IO-QOL-2000 index) | 2 years
  Impact of incontinence on quality of life. Scores are from 0 to 28. Slight impact in quality of life = 0-14. Higher impact in quality of life = 15-28.
Satisfaction with the treatment (Visual analogue scale.) | 2 years
  Visual analogue scale. Minimun values: 0, máximum values: 10. Higher score means a high satisfaction with the treatment received.
Duration of the response to treatment | 2 years
  the duration of the response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Álvaro Zapico-Goñi, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No